CLINICAL TRIAL: NCT00886496
Title: A Multi-Center Study of the Safety, Tolerability, Pharmacokinetics and Dose Escalation of Intravenous Recombinant Human Mannose-Binding-Lectin (rhMBL) in MBL Deficient Pediatric Hematology/Oncology Patients With Fever and Neutropenia
Brief Title: Recombinant Human Mannose-Binding Lectin (MBL) in Treating Young Patients With MBL Deficiency and Fever and Neutropenia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled. IND withdrawn.
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000523819; ENZON-EZN-2232-03; NCI-07-C-0027
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2007-08

CONDITIONS: Fever, Sweats, and Hot Flashes; Infection; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neutropenia; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; fever, sweats, and hot flashes; neutropenia; infection; recurrent childhood small noncleaved cell lymphoma; stage I and II childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III and IV childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood lymphoblastic lymphoma; stage I and II childhood lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III and IV childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; childhood Burkitt lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood grade III lymphomatoid granulomatosis; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III and IV childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Fever; Hot Flashes; Infections; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neutropenia; Burkitt Lymphoma; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating | interventions — Mannose-Binding Lectin

INTERVENTIONS:
Biological: recombinant human mannose-binding lectin

SUMMARY:
RATIONALE: Recombinant human mannose-binding lectin (MBL) may be effective in preventing infection in young patients with fever and neutropenia receiving chemotherapy for blood disease or cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of recombinant human mannose-binding lectin in treating young patients with MBL deficiency and fever and neutropenia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of recombinant human mannose-binding lectin (MBL) in pediatric patients with MBL deficiency and fever and neutropenia who are undergoing cytotoxic chemotherapy for hematological/oncological disease.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine the pharmacodynamic effect of this drug in these patients.
* Determine nonspecific activation of complement by in vivo determination of C3d complement activation in patients treated with this drug.
* Determine the ex-vivo activity of recombinant MBL in opsonization capacity of patients' sera to yeast and bacteria.
* Determine immunogenicity of this drug in these patients.
* Determine the incidence and duration of fever and breakthrough infections in patients treated with this drug.

OUTLINE: This is a non-randomized, multicenter, open-label, prospective, cohort study. Patients are assigned to 1 of 2 treatment groups.

* Group I: Patients receive low-dose recombinant human mannose-binding lectin (MBL) IV over 1 hour within 72 hours of onset of fever and neutropenia.
* Group II: Patients receive high-dose recombinant human MBL IV over 1 hour within 72 hours of onset of fever and neutropenia.

Patients undergo blood collection periodically during study for pharmacokinetic, pharmacodynamic, MBL immunogenicity, and opsonization/phagocytosis studies.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing cytologic chemotherapy for hematological/oncological disease
* Must meet all of the following criteria:

  * Documented mannose-binding lectin (MBL) levels < 300 ng/mm³ within the past week
  * Fever (oral temperature > 100.4° F)
  * Neutropenia, defined as absolute neutrophil count ≤ 1,000/mm³ with the anticipation that the counts will fall below 500/mm^3
  * Receiving broad spectrum antibiotic therapy for fever and neutropenia

PATIENT CHARACTERISTICS:

* No serious illness, in the opinion of the principal investigator, that would preclude study compliance
* No known allergic reactions to mannose-binding lectin or other human plasma products
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception during and for ≥ 30 days after completion of study treatment
* AST and ALT ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Creatinine clearance > 60 mL/min OR creatinine based on age as follows:

  * No more than 0.8 mg/dL (for patients 5 years of age and under)
  * No more than 1.0 mg/dL (for patients 6-9 years of age)
  * No more than 1.2 mg/dL (for patients 10-12 years of age)
  * No more than 1.4 mg/dL (for patients over 13 years of age [female])
  * No more than 1.5 mg/dL (for patients 13-15 years of age [male])
  * No more than 1.7 mg/dL (for patients of 16 years of age [male])
* No poor venous access that would preclude IV drug delivery or multiple blood draws
* Patients on hemodialysis must be able to tolerate IV fluid on non-dialysis days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since prior investigational agents

  * Investigational use of an FDA-approved drug allowed
* No concurrent preparative regimen for a bone marrow or hematopoietic stem cell transplantation
* No concurrent participation in another clinical trial with an investigational agent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-11; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Toxicity
Pharmacokinetics
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania